CLINICAL TRIAL: NCT02388178
Title: Assessment of 1450 Ppm Fluoride/Arginine Toothpaste Using an Intra-oral Remineralization-demineralization Model.
Brief Title: To Determine the Ability of a New Product Formulation to Remineralize an Early Caries Lesion by an In-situ Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to business reasons.
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ERO-2014-CAI-02-RPS
Record Dates: First submitted 2015-02-04; First posted 2015-03-13 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Amino Acids; Arginine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluoride free, silica based toothpaste (Placebo Comparator): Control toothpaste containing no anti-cavity ingredients
  Interventions: Drug: Control toothpaste containing no anti-cavity ingredients; Drug: Experimental toothpaste containing fluoride and amino acid (arginine); Drug: Fluoride toothpaste containing fluoride as the anti-cavity ingredient
- fluoride + amino acid in a silica toothpaste (Experimental): Experimental toothpaste containing fluoride and amino acid (arginine)
  Interventions: Drug: Control toothpaste containing no anti-cavity ingredients; Drug: Experimental toothpaste containing fluoride and amino acid (arginine); Drug: Fluoride toothpaste containing fluoride as the anti-cavity ingredient
- 1450 ppm fluoride in a silica base toothpaste (Active Comparator): Fluoride toothpaste containing fluoride as the anti-cavity ingredient
  Interventions: Drug: Control toothpaste containing no anti-cavity ingredients; Drug: Experimental toothpaste containing fluoride and amino acid (arginine); Drug: Fluoride toothpaste containing fluoride as the anti-cavity ingredient

INTERVENTIONS:
Drug: Control toothpaste containing no anti-cavity ingredients — Brush whole mouth with study toothpaste 2x/day for the 2 week test period. Each brushing routine is 1 minute whole mouth brushing with oral retainer in mouth, spit out toothpaste residue and wait for 1 minute before rinsing with water.
  Other Names: Fluoride free toothpaste control
Drug: Experimental toothpaste containing fluoride and amino acid (arginine) — Brush whole mouth with study toothpaste 2x/day for the 2 week test period. Each brushing routine is 1 minute whole mouth brushing with oral retainer in mouth, spit out toothpaste residue and wait for 1 minute before rinsing with water.
  Other Names: Experimental toothpaste
Drug: Fluoride toothpaste containing fluoride as the anti-cavity ingredient — Brush whole mouth with study toothpaste 2x/day for the 2 week test period. Each brushing routine is 1 minute whole mouth brushing with oral retainer in mouth, spit out toothpaste residue and wait for 1 minute before rinsing with water.
  Other Names: Fluoride only toothpaste control

SUMMARY:
This is a double blind, cross-over, controlled clinical trial utilizing thirty (30) adults to evaluate remineralization of early caries lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or female subjects 18 to 50 years inclusive
2. Minimum of 20 natural uncrowned teeth (excluding third molars) must be present
3. Willing to wear retainer 24 hours per day
4. No active, unrestored cavities
5. Have normal salivary flow rate (stimulated and unstimulated flow of ≥0.7 ml/min and ≥ 0.2 ml/min respectively) ascertained from a preliminary sialometry
6. Available throughout entire study
7. Willing to use only assigned products for oral hygiene throughout the duration of the study
8. Must give written informed consent
9. Must be in good general health
10. No known history of allergy to personal care/consumer products or their ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study

Exclusion Criteria:

1. Advanced periodontal disease
2. Medical condition which requires premedication prior to dental visits/procedures
3. Not enough teeth to secure the oral retainer
4. Diseases of the soft or hard oral tissues
5. Wear an Orthodontic appliances
6. Impaired salivary function
7. Current use drugs that can affect salivary flow
8. Use antibiotics one (1) month prior to or during this study
9. Pregnant or breastfeeding
10. Participate in another clinical study one (1) week prior to the start of the washout period or during this 9-week study period
11. Use tobacco products
12. Allergic to common toothpaste ingredients
13. Allergic to amino acids
14. Immune compromised individuals (HIV, AIDS, immuno-suppressive drug therapy)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Mineral Change (delta Z) | Baseline
  Tooth samples of human enamel are placed in a retainer and worn by each study subject. Enamel block samples will be x-rayed and analyzed for mineral level (volume % of micrometer of lesions , vol% µm) before being placed in the retainer. These baseline values will be compared with the post use delta mineral change (∆ Z).
Mineral Change (delta Z) | 2 weeks (from Baseline)
  Tooth samples of human enamel are placed in a retainer and worn by each study subject. After 2 weeks of wearing the study retainer, samples from the retainer will be x-rayed and analyzed for mineral level (volume % of micrometer of lesions , vol% µm). These post use values will be compared to the Baseline values to give a delta mineral change (∆ Z).

CONTACTS AND LOCATIONS:
Overall Officials: Bennet Amaechi, PhD, DDS, Principal Investigator — University of Texas